CLINICAL TRIAL: NCT05696912
Title: Resolving Unsolved Rare Diseases : Functional Tests and New Diagnosis Strategy to Study Genetic Variants From High-throughput Sequencing (RID)
Brief Title: Functional Tests to Resolve Unsolved Rare Diseases. Rares.
Acronym: RID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU BX 2021/40
Record Dates: First submitted 2022-12-07; First posted 2023-01-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Intellectual Disability; Rubinstein-Taybi Syndrome; Cystic Fibrosis; Congenital Heart Defect; Periventricular Nodular Heterotopia; Neurodegeneration With Brain Iron Accumulation (NBIA); Albinism
Keywords: Variant of unknown significance; Functional genetics; Translational research; RNAseq; Gene expression regulation
MeSH Terms: conditions — Intellectual Disability; Rubinstein-Taybi Syndrome; Cystic Fibrosis; Heart Defects, Congenital; Periventricular Nodular Heterotopia; Pantothenate Kinase-Associated Neurodegeneration; Albinism

STUDY DESIGN:
Intervention Model Description: Ex-vivo approach concerning 25 patients with blood sample in PAXgene tubes or skin biopsy and RNA-Seq analysis.
  In-vitro approach concerning 25 patients without specific samples needed for analysis in minigene or luciferase assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ex-vivo and In-vitro approach (Other): Ex-vivo approach concerning 25 patients with blood sample in PAXgene tubes or skin biopsy and RNA-Seq analysis.
  In-vitro approach concerning 25 patients without specific samples needed for analysis in minigene or luciferase assay
  Interventions: Genetic: Ex-vivo approach concerning 25 patients; Genetic: In-vitro approach concerning 25 patients

INTERVENTIONS:
Genetic: Ex-vivo approach concerning 25 patients — Ex-vivo approach concerning 25 patients with blood sample in PAXgene tubes or skin biopsy and RNA-Seq analysis
Genetic: In-vitro approach concerning 25 patients — In-vitro approach concerning 25 patients without specific samples needed for analysis in minigene or luciferase assay

SUMMARY:
Rares diseases are a heterogeneous group of conditions which need important tools for diagnosis.

The use of high-throughput sequencing is able to diagnose half of the patients. For the other part it is impossible to conclude due to the presence of variants of unknown significance (VOUS). Functional analysis are needed to bring strong argument to reclassify variants as pathogenic or benign. The main objective is to evaluate the diagnosis yield of this strategy.

DETAILED DESCRIPTION:
The main objective is the improvement of the diagnosis of rare genetic diseases. The investigator lab is expert for diagnosis of some rare diseases such as neurodevelopmental disorder, albinism, cystic fibrosis and congenital heart defect. Actually with implementation of high-throughput sequencing for diagnosis, a high number of genetic variants are found and need to be interpretated. The ACMG classification is used to classify variants with argument of variant frequency, predicted effect on protein and in-silico prediction. Functional evidence is a strong argument to help classify VOUS. The investigators propose the use of RNA-Seq, minigene and luciferase assay for study of VOUS to bring argument to classify them as benign or pathogenic.

ELIGIBILITY:
Inclusion Criteria:

* Minor and adult patient.
* Registered for the social security system.
* Informed consent signed by patient or parent of a minor patient.
* Patient affected by one of the rare diseases studied (albinism, congenital heart defect, cystic fibrosis, neurodevelopmental disease)
* Patient bearing variants of unknown significance (VOUS)

Exclusion Criteria:

* Refusal to participate in research protocol.
* Patient under administrative supervision
* Pregnant or nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of VOUS reclassified as pathogenic (class 5) or benign (class 1) | Inclusion visit
  It's the proportion of VOUS that could be definitively reclassified as pathogenic (class 5) or benign (class 1) according to the ACMG classification (Richards et al., 2015 and Appendix 1). Indeed currently only variants considered as pathogenic or probably pathogenic make it possible to confirm a diagnosis and to propose genetic offer genetic counseling to families and perform a prenatal diagnosis. This is an evaluation that will be carried out at the end of the analyses carried out

SECONDARY OUTCOMES:
Pre-analysis process : Time of sample transport to the laboratory | Inclusion visit
  Time of transport to the laboratory. To calculate this time, the time of collection and the time of receipt by the and the time of reception by the molecular genetics technician will be recorded
Pre-analysis process : Quality of RNA extraction (RNA Integrity Number, RIN) | Inclusion visit
  RNA quality measurement by RIN (RNA integrity number): very good >7, good >/=5, poor <5. Only RNA with RIN >5 will be retained.
Praticability :Characteristics and number of CPU (Central Processing Unit) | Inclusion visit
  Evaluation of bioinformatic ressources by measure of number of CPU needed and turnaround time for processing data
Praticability : Training time of Biologists for interpretation | Inclusion visit
  Evaluation of training time needed to interpret the data
Global cost | Inclusion visit
  Evaluation of cost of global analyse and each test

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MICHAUD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hopital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No